CLINICAL TRIAL: NCT05467410
Title: Optimal Timing of Computerized Cognitive Training for Older Intensive Care Unit Survivors
Acronym: OPTIMIZE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: American Association of Critical Care Nurses (Other)
Responsible Party: Principal Investigator, Maya Elias, PhD, RN, Assistant Professor, Department of Biobehavioral Nursing and Health Informatics, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00014922; 40067 (Other Grant/Funding Number: American Association of Critical-Care Nurses (AACN))
Record Dates: First submitted 2022-04-21; First posted 2022-07-20 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Critical Illness; Cognitive Impairment; Circadian Dysrhythmia; Intensive Care Unit Delirium; Aging; Older People
MeSH Terms: conditions — Critical Illness; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, experimental design
Who Masked: Outcomes Assessor
Masking Description: Study personnel evaluating cognitive function outcomes will use standardized cognitive measures and will be blinded to participants' group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COG-AM (Experimental): 30-minute morning session of a laptop-based computerized cognitive training intervention, delivered between the hours of 09:00 AM - 12:00 PM, in addition to UC
  Interventions: Behavioral: COG-AM
- COG-PM (Experimental): 30-minute afternoon/evening session of a laptop-based computerized cognitive training intervention, delivered between the hours of 15:00 PM - 18:00 PM, in addition to UC
  Interventions: Behavioral: COG-PM
- UC (No Intervention): Standard post-ICU inpatient care/usual care, which includes physical/occupational therapy as ordered by treatment team

INTERVENTIONS:
Behavioral: COG-AM — Participants who are randomized to the COG-AM intervention group will be asked to complete 30-minute computerized cognitive training (Lumosity cognitive training program) sessions during morning hours (between 09:00-12:00), for a total of 7 days or until hospital discharge, whichever comes first. Participants will complete cognitive training sessions in each of the following subdomains: memory, attention, problem solving, cognitive flexibility, and processing speed.
  Arms: COG-AM
Behavioral: COG-PM — Participants who are randomized to the COG-PM intervention group will be asked to complete 30-minute computerized cognitive training (Lumosity cognitive training program) sessions during late afternoon/early evening hours (between 15:00-18:00), for a total of 7 days or until hospital discharge, whichever comes first. Participants will complete cognitive training sessions in each of the following subdomains: memory, attention, problem solving, cognitive flexibility, and processing speed.
  Arms: COG-PM

SUMMARY:
More than 60% of intensive care unit (ICU) patients are adults ages 60 and older, who are at high risk for ICU-acquired cognitive impairment. After ICU discharge, ICU survivors often experience sleep disturbances and inactivity, and almost 80% of ICU patients experience disturbances in circadian rhythm, which may affect cognitive function. Understanding the optimal, chronotherapeutic timing of cognitive interventions is crucial to promote circadian realignment and cognitive function, and may improve intervention feasibility, acceptability, and efficacy. Specific Aim 1 will determine feasibility, acceptability, and preliminary effect sizes for: 1) a morning session of a computerized cognitive training intervention [COG]; and 2) a late afternoon/early evening session of the COG intervention; compared to 3) standard inpatient care/usual care [UC]. Specific Aim 2 will examine circadian rhythm parameters to determine the optimal timing of the daily COG intervention. Exploratory Aim 3 will explore if the effects of the COG intervention on cognitive function are mediated by daytime activity, and explore if selected biological and clinical factors moderate intervention effects on cognitive function.

DETAILED DESCRIPTION:
Over 60% of intensive care unit (ICU) patients are older adults (ages 60 and older). Up to 40% of ICU survivors experience cognitive impairment that is comparable in severity to moderate traumatic brain injury, while 25% have symptoms similar to mild Alzheimer's disease after hospital discharge. Older ICU survivors are at high risk for ICU-acquired cognitive impairment, often leading to a protracted recovery in a care facility. Several factors, including circadian misalignment (observed in about 75-80% of ICU patients), may decrease effects of interventions designed to improve cognitive function. Further, daytime activity is essential for recovery from critical illness and to promote circadian realignment, yet ICU survivors experience profound inactivity. The scientific premise of the proposed research is that identifying the optimal circadian timing of cognitive interventions for older ICU survivors may improve intervention feasibility, acceptability, and efficacy. Interventions targeting symptoms (i.e., disturbances in circadian rhythm and cognitive impairment) may deliver similar outcomes across conditions that require ICU admission (e.g., cancer, heart failure, pneumonia, hip fracture). To date, interventions have not been evaluated in older ICU survivors that simultaneously target circadian misalignment and cognitive impairment. Moreover, because circadian misalignment adversely affects cognitive function, understanding the optimal timing of cognitive interventions is crucial to promote both circadian realignment and cognitive function. Specific Aim 1 will determine feasibility, acceptability, and preliminary effect sizes for: 1) a morning session of a computerized cognitive training intervention [COG]; and 2) a late afternoon/early evening session of the COG intervention; compared to 3) standard inpatient care/usual care [UC]. Specific Aim 2 will examine circadian rhythm parameters to determine the optimal timing of the daily COG intervention. Exploratory Aim 3 will explore if the effects of the COG intervention on cognitive function are mediated by daytime activity, and explore if selected biological and clinical factors moderate intervention effects on cognitive function. The proposed early-stage clinical trial will be the first to evaluate chronotherapeutic timing of a computerized cognitive training intervention for hospitalized older ICU survivors after ICU discharge, to initiate early cognitive recovery on a post-ICU unit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years
* ICU length of stay ≥ 24 hours
* Active transfer order or expected discharge from ICU to a post-ICU unit
* Fluent in English
* Functional independence prior to hospital admission (Katz Index = 6)
* No suspicion of Alzheimer's disease/dementia
* Current hospitalization at University of Washington Medical Center or Harborview Medical Center

Exclusion Criteria:

* Documented history or suspicion of Alzheimer's disease/dementia, or current prescription of anti-dementia medication
* Documented history of bipolar disorder or schizophrenia
* Documented acute stroke or acute traumatic brain injury
* Severe visual impairment
* Severe hearing impairment
* Severe dominant arm paresis/paralysis
* Transfer from inpatient rehabilitation or skilled nursing care facility

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of morning-only sessions of computerized cognitive training | 7 days
  A retention rate of >70% will determine feasibility: the percentage of participants who complete at least 60 minutes of COG-AM sessions and all cognitive outcome assessments. Adherence to the COG-AM intervention will be defined as the proportion of minutes spent training by the total minutes required per protocol (total minutes trained / [30 minutes x number of intervention days]).
Feasibility of afternoon/evening-only sessions of computerized cognitive training | 7 days
  A retention rate of >70% will determine feasibility: the percentage of participants who complete at least 60 minutes of COG-PM sessions and all cognitive outcome assessments. Adherence to the COG-PM intervention will be defined as the proportion of minutes spent training by the total minutes required per protocol (total minutes trained / [30 minutes x number of intervention days]).
Acceptability of morning-only sessions of computerized cognitive training | 7 days
  Likert-type surveys including open-ended questions will be collected regarding acceptability of the COG-AM intervention. To evaluate tolerability, reasons why participants were unable to complete COG-AM sessions in their entirety will be recorded.
Acceptability of afternoon/evening-only sessions of computerized cognitive training | 7 days
  Likert-type surveys including open-ended questions will be collected regarding acceptability of the COG-PM intervention. To evaluate tolerability, reasons why participants were unable to complete COG-PM sessions in their entirety will be recorded.

SECONDARY OUTCOMES:
Cognitive function: global cognition | 7 days
  National Alzheimer's Coordinating Center Uniform Data Set: Montreal Cognitive Assessment; range: 0-30; higher scores indicate better performance
Cognitive function: verbal working memory | 7 days
  National Alzheimer's Coordinating Center Uniform Data Set: Number Span Test Forward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: executive function | 7 days
  National Alzheimer's Coordinating Center Uniform Data Set: Number Span Test Backward; number of correct trials, range: 0-14; higher scores indicate better performance
Cognitive function: set-shifting | 7 days
  National Alzheimer's Coordinating Center Uniform Data Set: Oral Trail Making Test; time in seconds, range: 0-300; higher scores indicate worse performance
Circadian rhythm of continuous body temperature | 7 days
  Circadian rhythm: amplitude, acrophase, mesor via continuous body temperature obtained from wearable sensors
Activity counts per minute | 7 days
  Daytime activity: activity counts per minute during daytime hours via wrist actigraphy
Total sleep time in minutes | 7 days
  Nighttime sleep: total sleep time in minutes during nighttime hours via wrist actigraphy

CONTACTS AND LOCATIONS:
Overall Officials: Maya N Elias, PhD, MA, RN, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington